CLINICAL TRIAL: NCT04948359
Title: Determining Optimal Cuff Volume for Cuffed Endotracheal Tubes Commonly Used in Pediatric Patients: a Prospective Observational Study
Brief Title: Determining Optimal Cuff Volume in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Kahir Güneş, Specialist physician, Ankara City Hospital Bilkent
Other Study IDs: E2-21-76
Record Dates: First submitted 2021-06-28; First posted 2021-07-01 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Cuff; Airway Edema; Children, Only; Tracheal Intubation Morbidity
Keywords: Airway ultrasound; Cuffed endotracheal tube; Cuff volume; Cuff pressure; Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I (The patients intubated with cuffed ETT of ID number 4.5): Groups are classified according to endotracheal tube ID numbers. In this group we aimed to determine the optimal cuff volume that ensures airway safety in pediatric patients intubated with a 4.5 size internal diameter (ID) endotracheal cuff tube.
  Interventions: Other: Group I (The patients intubated with cuffed ETT of ID number 4.5)
- Group II (The patients intubated with cuffed ETT of ID number 5.0): Groups are classified according to endotracheal tube ID numbers. In this group we aimed to determine the optimal cuff volume that ensures airway safety in pediatric patients intubated with a 5.0 size internal diameter (ID) endotracheal cuff tube.
  Interventions: Other: Group II (The patients intubated with cuffed ETT of ID number 5.0)
- Group III (The patients intubated with cuffed ETT of ID number 5.5): Groups are classified according to endotracheal tube ID numbers. In this group we aimed to determine the optimal cuff volume that ensures airway safety in pediatric patients intubated with a 5.5 size internal diameter (ID) endotracheal cuff tube.
  Interventions: Other: Group III ( The patients intubated with cuffed ETT of ID number 5.5)

INTERVENTIONS:
Other: Group I (The patients intubated with cuffed ETT of ID number 4.5) — Groups are classified according to endotracheal tube ID numbers. Inflating the endotracheal tube cuff with more than normal volume leads to decreased capillary blood flow and mucosal damage, while inflating the endotracheal tube cuff with less than normal volume leads to insufficient ventilation of the patient and an increase in the risk of pulmonary aspiration. The cuff pressure safety range is recommended between 20-30 cmH2O to prevent gas leakage and the risk of aspiration. We aimed to determine the optimal cuff volume that ensures airway safety in pediatric patients intubated with a 4.5 size inner diameter (ID) endotracheal cuff tube. Choosing the appropriate tube for endotracheal intubation is of great importance, especially in children. In our study, the transverse diameter of the subglottic airway will be measured by USG for the selection of the appropriate ETT to be used for each patient (the formulas for the selection of ETT in the literature will be used)
  Groups: Group I (The patients intubated with cuffed ETT of ID number 4.5)
Other: Group II (The patients intubated with cuffed ETT of ID number 5.0) — Groups are classified according to endotracheal tube ID numbers. Inflating the endotracheal tube cuff with more than normal volume leads to decreased capillary blood flow and mucosal damage, while inflating the endotracheal tube cuff with less than normal volume leads to insufficient ventilation of the patient and an increase in the risk of pulmonary aspiration. The cuff pressure safety range is recommended between 20-30 cmH2O to prevent gas leakage and the risk of aspiration. We aimed to determine the optimal cuff volume that ensures airway safety in pediatric patients intubated with a 5.0 size inner diameter (ID) endotracheal cuff tube. Choosing the appropriate tube for endotracheal intubation is of great importance, especially in children. In our study, the transverse diameter of the subglottic airway will be measured by USG for the selection of the appropriate ETT to be used for each patient (the formulas for the selection of ETT in the literature will be used)
  Groups: Group II (The patients intubated with cuffed ETT of ID number 5.0)
Other: Group III ( The patients intubated with cuffed ETT of ID number 5.5) — Groups are classified according to endotracheal tube ID numbers. Inflating the endotracheal tube cuff with more than normal volume leads to decreased capillary blood flow and mucosal damage, while inflating the endotracheal tube cuff with less than normal volume leads to insufficient ventilation of the patient and an increase in the risk of pulmonary aspiration. The cuff pressure safety range is recommended between 20-30 cmH2O to prevent gas leakage and the risk of aspiration. We aimed to determine the optimal cuff volume that ensures airway safety in pediatric patients intubated with a 5.5 size inner diameter (ID) endotracheal cuff tube. Choosing the appropriate tube for endotracheal intubation is of great importance, especially in children. In our study, the transverse diameter of the subglottic airway will be measured by USG for the selection of the appropriate ETT to be used for each patient (the formulas for the selection of ETT in the literature will be used)
  Groups: Group III (The patients intubated with cuffed ETT of ID number 5.5)

SUMMARY:
Background and Aim: Cuffed endotracheal tubes with appropriate size, good cuff design and cuff pressure monitoring in pediatric patients can be used safely without increasing airway morbidity. Inflating the endotracheal tube cuff with more than normal volume may lead to decreased capillary blood flow and mucosal damage, while inflating the endotracheal tube cuff with less than normal volume may lead to an increase in the risk of inadequate ventilation and pulmonary aspiration. In this study, we aimed to determine an optimal cuff inflation volume to achieve safe cuff pressure (20-25 cm H2O) in cuffed endotracheal tubes with an inner diameter of 4.5, 5.0, 5.5 mm, which are commonly used in pediatric anesthesia clinical practice.

DETAILED DESCRIPTION:
Design:

This is a prospective, single blinded, observational study. In case of 2 independent variables in the multiple linear regression analysis, the required sample size was calculated as at least 40 in order to determine the large effect width (f2=0.35) at 0.80 power and 0.05 error levels. Since the study will be carried out with 3 different tube diameters, the sample size has been determined as 120 in total (G*Power software 3.1.9). In the Bland and Altman method, it was stated that when there are at least 100 observations, the 95% confidence level can be determined in the range of ±0.34s (where "s" is the standard deviation of the differences between the two measurements). For this reason, it is seen that the determined sample number of 120 is also sufficient for the Bland&Altman method. Power analysis was made with G*Power 3.1.9.7 statistical package program; group=3, n=127 (n1=42, n2=43, n3=42), α=0.05, Effect Size (f)=0.34; power = 93%.

Methods: Pediatric patients younger than 18 yr old who will be operated in our hospital and intubated with cuffed tubes numbered 4.5, 5.0, and 5.5 under general anesthesia will be included in this prospective observational study. After standard monitoring in the supine position, anesthesia will be induced with a mixture of O2 / air (50/50%) and 8% Sevoflurane, and then vascular access will be established. Intravenous (IV) 2-3 mg/kg propofol and 1 μgr/kg fentanyl will be administered to patients with IV access. For muscle relaxation after loss of consciousness, 0.5 mg/kg rocuronium will be given IV. After the patients are paralyzed, a 3 cm roll pad will be placed under their shoulders and airway ultrasonography imaging will be performed with the head slightly extended and in the supine-neutral position. The linear probe will be placed transversely in the anterior neck of the patients and moved in a cefo-caudal direction to view the cricoid cartilage. The cricoid cartilage appears as a hypoechoic round structure with hyperechoic margins. At this level, the transverse diameter of the subglottic air column will be measured in millimeters (mm) on the USG image. The formulas in the literature and the subglottic transverse trachea diameter measured by ultrasound will be used to select the most appropriate endotracheal tube for the pediatric patients. After the appropriate cuffed tube is attached to the patient, the cuff will be inflated with air through a 5 milliliter (ml) injector, and cuff pressure will be measured with a cuff manometer. The optimal cuff volume will be determined by giving or withdrawing the 0.2 ml volume to ensure optimum cuff pressure (20-25 cmH2O) and this value will be recorded. Demographic data of the patients, subglottic transverse airway diameter measured by ultrasonography, endotracheal tube number placed in the patient, given cuff volume, measured cuff pressure value, tube change requirement, peak airway pressure, operation time and postoperative airway complications (sore throat, desaturation, stridor, hoarseness, cough) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients younger than 18 yr old who will be operated in our hospital and intubated with cuffed tubes numbered 4.5, 5.0, and 5.5 under general anesthesia are included in this study.

Exclusion Criteria:

* ASA physical status score of III and IV,
* Tracheostomy, airway obstruction or other airway anatomical abnormalities,
* Difficult intubation prediction,
* History of airway hyperreactivity or bronchial asthma,
* Body mass index above the 85th percentile and below the 5th percentile,
* Patients whose parents were unable to read, understand and sign the consent form or whose parents did not want to sign the consent form will not included in the study.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients younger than 18 yr old who will be operated in our hospital and intubated with cuffed tubes numbered 4.5, 5.0, and 5.5 under general anesthesia
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Optimal intracuff volume | during surgery
  To obtain the minimum and optimal cuff volume that will provide adequate ventilation and protect from pulmonary aspiration in pediatric patients who is intubated with cuffed endotracheal tubes inner diameter of 4.5, 5.0, 5.5 mm.
Formula for optimal cuff volume. | 15 minute
  We would like to create a formula to calculate the estimated cuff volume that should be inflated within the safe cuff pressure range for each patient intubated with an ETT ID number 4.5, 5.0, and 5.5.

SECONDARY OUTCOMES:
Formula for subglottic transverse tracheal diameter | 15 minute
  We would like to develop a formula to predict subglottic transverse tracheal diameter with a regression model to be established by usin subglottic tracheal diameter data measured by USG in each patient.
Postoperative complications | 1 hour
  The other secondary objective of this study is to examine correlation between cuff volume and postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Kahir Güneş, Principal Investigator — Ankara City Hospital Bilkent; Sengül Özmert, Study Director — Ankara City Hospital Bilkent; Feyza Sever, Study Director — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Çankaya, Turkey (Türkiye)

REFERENCES:
- [Derived] Gunes K, Sever F, Ozmert S. Determining optimal cuff volume for cuffed endotracheal tubes commonly used in pediatric patients: A prospective observational study. Saudi Med J. 2024 Feb;45(2):147-153. doi: 10.15537/smj.2024.45.2.20230578. PMID 38309733